CLINICAL TRIAL: NCT02356666
Title: Prevalence of Nocturnal Hypoventilation in Neuromuscular Diseases According to Different Definitions
Acronym: TcCO2
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: 1817118
Record Dates: First submitted 2014-12-17; First posted 2015-02-05 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Neuromuscular Disease
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Different definitions of nocturnal hypoventilation are used in the recent literature. The investigators aimed to compare the prevalence of nocturnal hypoventilation in a neuromuscular disease's population according to different definitions issued from the literature.

DETAILED DESCRIPTION:
Different definitions of nocturnal hypoventilation are used in the recent literature. Basing on retrospective data review, we aimed to compare the prevalence of nocturnal hypoventilation in the cohort of neuromuscular disease's patients followed at our reference center, according to different definitions issued from the literature.

ELIGIBILITY:
Inclusion Criteria:

* Neuromuscular disease
* Age ≥18 years
* Non mechanically ventilated

Exclusion Criteria:

* Long-term oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuromuscular disease
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Differences in the prevalence of nocturnal hypoventilation according to different previously proposed definitions | Baseline (Day 1)
  The prevalence of nocturnal hypoventilation (percentage of patients diagnosed as having hypoventilation over the total population) according to the different definition available in the literature will be described

SECONDARY OUTCOMES:
Concordance between the diagnostic criteria | Baseline (Day 1)
  Concordance between the different diagnostic criteria of hypoventilation
sensibility/specificity of the different criteria to identify daytime alveolar hypoventilation (defined on blood gas analysis) | Baseine (Day 1)
  sensibility/specificity of the different criteria to identify daytime alveolar hypoventilation (defined on blood gas analysis)
Prognostic value of the different definitions of nocturnal hypoventilation | 5 years
  The ability of the examined definition to predict the need for mechanical ventilation will be investigated, defined as appearance of daytime hypercapnia or beginning of mechanical ventilation and/or mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Ogna, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France